CLINICAL TRIAL: NCT07400965
Title: Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel Group Phase 2 Trial Evaluating the Safety and Efficacy of GLK-321 in Subjects With Demodex Blepharitis
Brief Title: Randomized, Placebo-controlled Trial Evaluating the Safety and Efficacy of GLK-321 in Subjects With Demodex Blepharitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-321-01
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Demodex Blepharitis
Keywords: demodex blepharitis
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- GLK-321 low dose BID (Experimental): Low dose of GLK-321 administered twice daily (BID) to both eyes
  Interventions: Drug: GLK-321 low dose BID
- GLK-321 mid dose BID (Experimental): Mid dose of GLK-321 administered twice daily (BID) to both eyes
  Interventions: Drug: GLK-321 mid dose BID
- GLK-321 high dose BID (Experimental): High dose of GLK-321 administered twice daily (BID) to both eyes
  Interventions: Drug: GLK-321 high dose BID
- GLK-321 high dose QD (Experimental): High dose of GLK-321 administered once daily (QD) to both eyes
  Interventions: Drug: GLK-321 high dose QD
- Placebo BID (Placebo Comparator): Placebo administered twice daily (BID) to both eyes
  Interventions: Drug: Placebo BID

INTERVENTIONS:
Drug: GLK-321 low dose BID — Twice daily administration of low dose GLK-321 to both eyes
  Arms: GLK-321 low dose BID
Drug: GLK-321 mid dose BID — Twice daily administration of mid dose GLK-321 to both eyes
  Arms: GLK-321 mid dose BID
Drug: GLK-321 high dose BID — Twice daily administration of high dose GLK-321 to both eyes
  Arms: GLK-321 high dose BID
Drug: GLK-321 high dose QD — Once daily administration of high dose GLK-321 to both eyes
  Arms: GLK-321 high dose QD
Drug: Placebo BID — Twice daily administration of placebo to both eyes
  Arms: Placebo BID

SUMMARY:
This is a randomized, double-masked, placebo-controlled, dose-ranging, parallel-group, multi-center study designed to evaluate the safety and efficacy of GLK-321 in patients with Demodex blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* Signs of Demodex blepharitis in at least one eye
* Best Spectacle Corrected Visual Acuity (BSCVA) of 20/80 Snellen or better in each eye

Exclusion Criteria:

* Presence of eczema or dermatitis in the ocular region of either eye
* Use of lid hygiene products within 14 days of Screening
* Active ocular infection or inflammation, other than blepharitis, in either eye at Screening
* Women who are pregnant, planning a pregnancy, or nursing
* Have used an investigational drug or device within 30 days prior to Screening or concurrently enrolled in another investigational drug or device trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of study eyes with elimination of collarettes | 6 weeks
  Percentage of study eyes that had eyelash collarettes due to Demodex blepharitis at the onset of treatment who demonstrate absence of collarettes after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, MD, Study Director — Glaukos Corporation
Locations (1):
- Glaukos Clinical Study Site, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No